CLINICAL TRIAL: NCT01683955
Title: Topical Tranexamic Acid and Acute Blood Loss in Total Hip Arthroplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TEAHIPS
Record Dates: First submitted 2012-09-08; First posted 2012-09-12 (Estimated); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Acute Blood Loss Anemia; Osteoarthritis, Hip
Keywords: Tranexamic Acid; Blood transfusion; Total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic Acid (Experimental): Topical tranexamic acid (2g/100mL) applied during unilateral total hip arthroplasty.
  Interventions: Drug: Tranexamic acid
- Placebo (Placebo Comparator): 100mL 0.9% sterile saline, applied topically
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Topical tranexamic acid (2g/100mL 0.9% saline)
  Other Names: cyclokapron
  Arms: Tranexamic Acid
Drug: Placebo — 100mL 0.9% sterile saline
  Arms: Placebo

SUMMARY:
This study aims to assess postoperative blood loss and transfusion rates in total hip replacement after one-time administration of topical tranexamic acid.

DETAILED DESCRIPTION:
Autologous (donor) blood transfusion is an expensive and common occurrence after total hip replacement. There have been many proposed adjunctive measures to decrease intraoperative and postoperative blood loss during such surgery. Most of these include thrombin inhibition, so-called "minimally- invasive" techniques or instrumentation, or other adjunctive drugs. Hitherto, tranexamic acid, a specific drug that promotes part of the clotting cascade, has been used extensively in multiple areas of surgery with multiple studies evaluating its efficacy in cardiac surgery, spinal procedures, and as a dental swishing solution after tooth extraction. There have been small studies evaluating intravenous tranexamic acid and its effect on total hip replacements, with some promising results. The topical form of TA has been evaluated in only one prospective, randomized clinical trial with a significant decrease in postoperative blood loss and a trend towards decreased autologous blood transfusion rates. This study proposes to further evaluate tranexamic acid as an inexpensive and viable option for use in total hip arthroplasty. The topical form of the drug has been shown to achieve these hemostatic effects without increasing the risk of blood clots after surgery. A rigorous analysis of the effects of tranexamic acid demand a more standardized approach. Such a regimen is practiced at Henry Ford Hospital as all patients on the Adult Reconstruction service are placed on an identical dose of enoxaparin (a subcutaneous blood thinner) postoperatively for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients over age eighteen
* Primary unilateral total hip arthroplasty at Henry Ford Hospital (Detroit, Michigan, United States) and Henry Ford West Bloomfield Hospital (West Bloomfield, Michigan, United States)

Exclusion Criteria:

* patient history of venous thromboembolic disease or coagulopathy
* use of anticoagulant medications within 7 days of surgery
* history of arterial embolic disease
* history of Class III or IV heart failure
* renal failure
* intraoperative cardiovascular, pulmonary, orthopaedic, or anesthetic complication (MI, intraoperative fracture, vasopressor support, emergent intubation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2013-11-03 (Actual); Study Completion 2013-11-03 (Actual)

PRIMARY OUTCOMES:
postoperative blood loss | participants will be followed for the duration of hospital stay, an expected average of 3 days
  Preoperative and lowest postoperative hemoglobin

SECONDARY OUTCOMES:
postoperative transfusion rate | participants will be followed for the duration of hospital stay, an expected average of 3 days
  number of units transfused postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Michael Laker, M.D., Principal Investigator — Henry Ford Health Systems
Locations (2):
- United States (2):
  - Henry Ford Hospital, Detroit, Michigan
  - HFH Main campus, Detroit, Michigan